CLINICAL TRIAL: NCT00875849
Title: Phase II Study Evaluating Radiotherapy-chemotherapy and Cetuximab in Patients With Histologically Proven Squamous Cell Carcinoma of the Oral Cavity, Oropharynx, Hypopharynx, or Larynx and With a Poor Prognosis After Complete Surgical Resection
Brief Title: Chemotherapy, Radiation Therapy, and Cetuximab in Treating Patients With the Head and Neck Cancer
Acronym: AACER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/23; MERCK-CALACASS-AACER (Other Grant/Funding Number: MERCK); INCA-RECF0623 (Registry Identifier: INCA); 2007-004384-22 (EudraCT Number)
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2012-08

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cetuximab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Experimental)
  Interventions: Biological: cetuximab; Drug: cisplatin; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving chemotherapy together with radiation therapy and cetuximab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well chemotherapy given together with radiation therapy and cetuximab works in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate disease-free survival at 2 years in patients with poor prognosis squamous cell carcinoma of the head and neck treated with chemoradiotherapy and cetuximab after complete surgical resection.

Secondary

* Evaluate quality of life.
* Evaluate tolerability.
* Evaluate overall survival.
* Analyze germinal polymorphisms.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV on day 1. Treatment with cetuximab repeats every week for up to 8 courses. Patients also receive cisplatin IV on day 8. Treatment with cisplatin repeats every 3 weeks for up to 3 courses. Patients undergo concurrent radiotherapy 5 times a week for 7 weeks beginning on day 8.

After completion of study treatment, patients are followed at 1 month and then every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx
* Must have undergone complete macroscopic resection
* Presence of ≥ 1 of the following poor prognostic factors after complete resection:

  * Incomplete microscopic resection and N+
  * Complete microscopic resection and > 2 N+
  * Vascular and/or lymphatic embolism
  * At least 2 peripheral nerve invasions
  * Positive surgical margins and pT4 lesion
* No metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9 g/dL
* Bilirubin < 1.5 times upper limit of normal (ULN)
* Serum creatinine < 1.25 times ULN and/or creatinine clearance > 55 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No serious and disabling cardiac, renal, hepatic, or respiratory failure
* No coronary artery disease or myocardial infarction within the past year
* No uncontrolled cardiac arrhythmia
* Other active and serious diseases allowed at discretion of the investigator
* No known severe allergy to cisplatin, cetuximab, or any of their excipients
* No other malignant disease diagnosed within the past 5 years except for basal cell carcinoma of the skin or in situ cervical cancer
* No psychological, familial, social, or geographic situations that preclude clinical follow up

PRIOR CONCURRENT THERAPY:

* No prior treatment (except surgery) for this cancer or another head and neck cancer
* At least 3 months since prior treatment with an investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival at 2 years | 2 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Follana, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France